CLINICAL TRIAL: NCT06832293
Title: Measuring MS Symptoms in Relation to Menstrual Cycles: Exploring How MS Symptoms May be Affected at Different Times During a Menstrual Cycle in Females Living With Multiple Sclerosis
Brief Title: My MS and My Menstrual Cycle
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00140591
Record Dates: First submitted 2025-02-06; First posted 2025-02-18 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis; Menstrual Cycle
Keywords: Multiple Sclerosis; Menstrual Cycle; MS Symptoms; Fatigue; Cognition
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to understand how MS symptoms change during different phases of the menstrual cycle in individuals who menstruate living with MS (Multiple Sclerosis).

The main questions it aims to answer are:

1. Does fatigue get worse during certain phases of the menstrual cycle?
2. How do symptoms like thinking skills, pain, and mobility change throughout the cycle?

Participants will:

* Use the My Normative app to track their menstrual cycle and MS symptoms.
* Complete symptom check-ins at five points during their cycle for six months.
* Answer questions about fatigue, thinking skills, mood, sleep, and other MS symptoms at the start and end of the study.

These findings may help researchers better understand MS symptom patterns and improve symptom management.

ELIGIBILITY:
Inclusion Criteria:

* Female participants diagnosed with MS based on the 2024 McDonald Diagnostic criteria (biologically sex-based, any gender as long as not on hormonal gender-enhancing therapy)
* Aged 16 or older
* Experiencing menstruation with cycles ranging from 21 to 35 days
* Have entered menarche, still experiencing menstrual cycles, and have not yet entered menopause
* May be using hormonal contraceptive methods (e.g., oral contraceptives or hormonal IUDs)
* Able to speak English
* Willing to provide informed consent (mature minors will be assessed by their physician for consent eligibility)
* Able to complete questionnaires and operate the app

Exclusion Criteria:

* Diagnosed with CNS inflammation disorders other than MS, such as:

NMOSD (Neuromyelitis Optica Spectrum Disorder) or MOGAD (Myelin Oligodendrocyte Glycoprotein Antibody-associated Disease)

* Male or intersex individuals, given the inclusion criteria of requiring a uterus
* Females under 15 years of age
* Females who have not started menstruation
* Females who have stopped menstruation due to menopause or hysterectomy
* Pregnant or postpartum individuals within one year of delivery,
* Individuals currently breastfeeding
* Unable to provide informed consent, or not deemed a mature minor
* Unable to complete questionnaires and operate the app

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be female individuals with confirmed diagnosis of Multiple Sclerosis (MS) who experience a regular menstrual cycle.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Difference in the Modified Fatigue Impact Scale-5 (MFIS-5) Score Across Menstrual Cycle Phases Over Six Months | The MFIS-5 is assessed at baseline (study entry), five key points (menstrual phases) throughout the participant's menstrual cycle every month for 6 months, and study completion (on average, 6 months later)
  The Modified Fatigue Impact Scale-5 (MFIS-5) measures the impact of fatigue on cognitive, physical, and psychosocial functions. It uses a 5-point Likert scale for each item, with the following scoring range for each of the 5 items:
  0: Never
  1. Rarely
  2. Sometimes
  3. Often
  4. Almost Always The total score is the sum of the five items, with a range from 0 to 20. A higher score indicates a greater impact of fatigue on daily functioning.
  In terms of interpreting the score:
  A score of 0 would indicate no impact from fatigue. A score of 20 would indicate the maximum possible impact of fatigue on daily functioning.
  This scale is used to assess fatigue severity in individuals with multiple sclerosis (MS) and other conditions where fatigue is a prominent symptom. A higher score reflects a greater degree of fatigue-related disruption to cognitive, physical, and social tasks.

SECONDARY OUTCOMES:
Qualitative Self-Reported Differences in Self-Perceived Cognitive Function Across Menstrual Cycle Phases | The Cognition Likert Scale is assessed at baseline (study entry) and at five key points (menstrual phases) throughout the participant's menstrual cycle every month for 6 months
  The Cognition Likert Scale measures self-perceived cognitive function in individuals with MS. It consists of two items rated on a 7-point Likert scale:
  1. Perceived Cognitive Function Compared to Peers (ex. 1 = Severely worse, 4 = Unchanged, 7 = Significantly better).
  2. Frequency of Cognitive Difficulties (ex. 1 = Never, 4 = Sometimes, 7 = All the time).
  Each item is interpreted independently.
  Interpreting the Score:
  A lower score on the Perceived Cognitive Function scale (e.g., 1-3) suggests greater cognitive impairment, while a higher score (e.g., 5-7) indicates better cognitive function compared to peers.
  A lower score on the Frequency of Cognitive Difficulties scale (e.g., 1-3) suggests fewer cognitive challenges, while a higher score (e.g., 5-7) indicates more frequent cognitive difficulties.
  This scale is used to assess cognitive function in individuals with MS, allowing for the identification of self-reported changes in cognition over time.
Qualitative Self-Reported Differences in Hospital Anxiety and Depression Scale (HADS) Scores | The HADS is assessed at baseline (study entry) and study completion (on average, 6 months later)
  The Hospital Anxiety and Depression Scale (HADS) measures symptoms of anxiety and depression in individuals with MS. It consists of 14 self-reported items, with 7 items assessing anxiety and 7 items assessing depression over the past week.
  Each item is rated on a 4-point Likert scale (0-3), with total scores ranging from 0 to 21 for anxiety and 0 to 21 for depression.
  Interpreting the Score:
  0-7: Normal (no significant symptoms) 8-10: Borderline anxiety or depression 11-21: Clinical levels of anxiety or depression Higher scores indicate greater severity of anxiety and/or depression symptoms. The HADS is widely used in clinical and research settings to assess emotional well-being in individuals with chronic conditions like MS.
Qualitative Self-Reported Difference in Mini-COPE Scores Across Menstrual Cycle Phases | The Mini-COPE is assessed at baseline (study entry), five key points (menstrual phases) throughout the participant's menstrual cycle every month for 6 months, and study completion (on average, 6 months later)
  The Mini-COPE (MS-Specific Brief COPE) measures coping strategies used in response to stress. The scale assesses problem-focused coping, emotion-focused coping, and maladaptive coping. It consists of 28 self-reported items, each rated on a 4-point
  Likert scale:
  0 = I hardly ever do this
  1. = I rarely do this
  2. = I do this often
  3. = I almost always do this
  Interpreting the Score:
  * Higher scores indicate more frequent use of a specific coping strategy.
  * Individual scores provide insight into which coping mechanisms are most commonly used in response to stress.
  The Mini-COPE is widely used in MS research to understand coping behaviors and their impact on psychological well-being.
Qualitative Self-Reported Difference in MFC (Motivation for Cognition) Scores Across Menstrual Cycle Phases | The MFC is assessed at baseline (study entry), five key points (menstrual phases) throughout the participant's menstrual cycle every month for 6 months, and study completion (on average, 6 months later)
  The Motivation for Cognition (MFC) Scale measures an individual's motivation to engage in cognitive tasks at a given moment. It consists of 10 self-reported items, each rated on a 7-point Likert scale:
  * 3 = Very strongly does not apply to me
  * 2 = Strongly does not apply to me
  * 1 = Somewhat does not apply to me 0 = Neutral
    * 1 = Somewhat applies to me
    * 2 = Strongly applies to me
    * 3 = Very strongly applies to me
  Interpreting the Score:
  * Higher scores indicate greater motivation for engaging in cognitive tasks.
  * Lower scores suggest reduced interest in or avoidance of cognitively demanding activities.
  The MFC Scale will be used to evaluate fluctuations in cognitive motivation over time, particularly in relation to MS symptoms and menstrual cycle phases.
Qualitative Self-Reported Difference in SymptoMScreen Scores Across Menstrual Cycle Phases | The SymptoMScreen is assessed at baseline (study entry), five key points (menstrual phases) throughout the participant's menstrual cycle every month for 6 months, and study completion (on average, 6 months later)
  The SymptoMSScreen measures the impact of MS symptoms on daily life and the accommodations individuals make due to these symptoms. The scale evaluates walking, hand function, spasticity, pain, sensory symptoms, bladder control, fatigue, vision, dizziness, cognition, depression, and anxiety. It consists of 12 self-reported items, each rated on a 7-point Likert scale:
  0 = No effect at all
  1. = Very mild limitation
  2. = Mild limitation
  3. = Moderate limitation
  4. = Severe limitation
  5. = Very severe limitation
  6. = Total limitation
  Interpreting the Score:
  - Higher scores indicate greater MS-related disability and symptom burden.
  The SymptoMSScreen is used in MS research to assess symptom severity and it's impact on daily functioning. It's use will help track symptom progression and variability across menstrual cycle phases.
Qualitative Self-Reported MSNQ (Multiple Sclerosis Neuropsychological Screening Questionnaire) Scores | The MSNQ will be assessed at baseline (study entry) and study completion (on average, 6 months later)
  The Multiple Sclerosis Neuropsychological Screening Questionnaire - Patient Version (MSNQ) assesses cognitive and emotional difficulties in individuals with MS. The scale assesses attention, memory, problem-solving, impulse control, and emotional regulation. It consists of 15 self-reported items, each rated on a 5-point Likert scale based on frequency and severity over the past three months:
  0 = Never, does not occur
  1. = Very rarely, no problem
  2. = Occasionally, seldom a problem
  3. = Quite often, interferes with life
  4. = Very often, very disruptive
  Interpreting the Score:
  - Higher scores indicate greater cognitive and emotional impairment related to MS.
  The MSNQ is commonly used in MS research to identify cognitive difficulties and their impact on daily life. The use of MSNQ will help track cognitive fluctuations across menstrual cycle phases.

CONTACTS AND LOCATIONS:
Overall Officials: Penny Smyth, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT06832293/Prot_SAP_002.pdf
  • Informed Consent Form (2024-10-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT06832293/ICF_001.pdf